CLINICAL TRIAL: NCT05624489
Title: Personalized Digital Behavior Change Interventions to Promote Oral Health
Brief Title: Micro-Randomized Trial to Optimize Digital Oral Health Behavior Change Interventions
Acronym: DCBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Vivek Shetty, DDS, DMD, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB#21-001471; UG3DE028723 (NIH)
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Dental Diseases
Keywords: Dental disease; Health Behavior Change; Oral Self Care Behaviors
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: Each participant-time point (which will occur twice daily, in the morning and the evening) will be randomized between a prompt containing an engagement strategy vs. no prompt.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Each participant-time point will be randomized between a prompt containing an engagement strategy vs. no prompt. A Bayesian algorithm will iteratively adjust the probability of receiving a prompt or no prompt at any time point, using brushing behavior data. Patterns suggesting positive effects of the prompts on brushing adherence will result in higher subsequent probabilities of receiving the prompts, whereas patterns suggesting null or negative effects will result in lower probabilities of receiving the prompts. A participant is assigned to an engagement prompt will be randomized equally between the three types of engagement strategies: (1) Standard reciprocity prompt: delivering non-contingent reward points as a "gift" to support goals; (2) Reciprocity by proxy prompt: delivering a message indicating a donation to the person's selected charity; (3) Curiosity prompt: delivering oral health information in a manner that motivates the participant to seek new knowledge and information.
  Interventions: Behavioral: Engagement Strategies

INTERVENTIONS:
Behavioral: Engagement Strategies — The study's mobile app (Oralytics) will be used to deliver engagement prompts. The prompts contain messages that leverage three engagement strategies: reciprocity, reciprocity by proxy, and curiosity.

SUMMARY:
The study will involve a 10-week Micro-Randomized Trial (MRT) to inform the delivery of prompts (via mobile app push notifications) designed to facilitate adherence to an ideal tooth brushing protocol (2x2x4; 2 sessions daily, 2 minutes per session, all 4 quadrants).

DETAILED DESCRIPTION:
The goal of the MRT is to investigate whether delivering (vs. not delivering) a prompt that contains engagement strategies grounded in decision science is beneficial in terms of promoting proximal oral health behavior (OHB) score, which reflects adherence to the 2x2x4 brushing protocol (Primary Aim) and also mobile health engagement (mHealth; Secondary Aim). Additionally, Exploratory Aims will concern (a) comparing different types of prompts in terms of proximal OHB score and mHealth engagement, (b) investigating the conditions in which prompts should be delivered to most effectively promote proximal OHB and mHealth engagement; and (c) investigating whether the effect of the engagement prompts (vs. no prompt) on OHB score varies across components of the 2x2x4 brushing regimen (i.e., frequency, duration, or coverage).

Participants will receive an electronic toothbrush (eBrush) and a mobile app (Oralytics) that contains well-established behavior change strategies (e.g., goal setting, monitoring adherence, and feedback). Participants will be randomized twice per day - in the morning and the evening - to receive either (a) a push notification containing one of three (randomly selected) engagement strategies or (b) no notification.

During the 10 weeks of the study, a Bayesian algorithm will iteratively adjust the probability of receiving a prompt or no prompt in any given randomization window, using prior behavioral data collected through the eBrush and mobile app. Data patterns suggesting positive effects of the prompts on adherence to brushing protocol, especially duration, will result in higher subsequent probabilities of receiving the prompts, whereas patterns suggesting null or negative effects will result in lower probabilities of receiving the prompts.

Study results will inform the implementation of a smartphone-delivered behavior change intervention that further adapts the delivery of engagement prompts based on passively collected information from an eBrush and the mobile app.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 or older.
* Fluent in English
* Dentulous/partially edentulous (18+ teeth; at least 2 teeth in each quadrant)
* Possess a smartphone (iOS or Android) with a data plan.
* Willing to allow the passive collection of data on tooth-brushing activities in the home setting for 10 weeks.

Exclusion Criteria:

* Not fluent in English
* Edentulous
* Unable to use a mobile device due to cognitive or physical impairments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Proximal adherence to 2x2x4 OHB | 24 hours
  Change in proximal OHB score between the current and next randomization

SECONDARY OUTCOMES:
Proximal mHealth engagement | 24 hours
  Engagement with Oralytics app (i.e., accessing the Oralytics app or clicking on the push notification) between the current and next randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Shetty, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be generated and made available to the research community. The dataset will be stripped of all codes or any other information that could be linked back to the original data or an individual participant. Prospective users of this dataset must agree to a confidentiality agreement and get permission from the Primary Investigator to use or share the data with anyone else. All external requests for data will be directed to Dr. Vivek Shetty. Prospective investigators will submit a written proposal to the PI outlining the question they will investigate, the specific variables that they need to answer that question, their analytic plan for answering that question, and documentation of sufficient Institutional Review Board oversight (e.g., approval or exemption). Investigators will also need to sign a confidentiality agreement.
Supporting Information: Study Protocol, CSR
Time Frame: 12 months after publication of primary analyses.
Access Criteria: All external requests for data will be directed to the PI (Dr. Vivek Shetty). Prospective investigators will submit a written proposal to the PI outlining the question they will investigate, the specific variables that they need to answer that question, their analytic plan for answering that question, and documentation of sufficient Institutional Review Board oversight (e.g., approval or exemption). Investigators will also need to sign a confidentiality agreement.

REFERENCES:
- [Background] Nahum-Shani I, Greer ZM, Trella AL, Zhang KW, Carpenter SM, Runger D, Elashoff D, Murphy SA, Shetty V. Optimizing an adaptive digital oral health intervention for promoting oral self-care behaviors: Micro-randomized trial protocol. Contemp Clin Trials. 2024 Apr;139:107464. doi: 10.1016/j.cct.2024.107464. Epub 2024 Feb 1. PMID 38307224